CLINICAL TRIAL: NCT06238583
Title: Copanlisib Expanded Access Program (EAP) for Patients Who, in the Opinion of Their Healthcare Provider, Are Deriving Benefit From Copanlisib Therapy
Brief Title: Expanded Access to Provide Copanlisib for Patients With Cancer Who Are Experiencing a Positive Response, as Determined by Their Doctors
Status: No longer available | Type: Expanded Access
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22702
Record Dates: First submitted 2024-01-24; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — copanlisib

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Copanlisib (Aliqopa, BAY80-6946) — Copanlisib is supplied as lyophilized preparation in a 6 mL injection vial. The total amount of copanlisib per vial is 60 mg. The recommended dose of copanlisib is 60 mg administered as a 1 hour intravenous (IV) infusion on Days 1, 8, and 15 of a 28-day treatment cycle on an intermittent schedule (3 weeks on and 1 week off), OR at a lower dose if dose reduction has occurred on prior treatment. Patients currently included on study protocols may continue their treatment regimen at the discretion of their healthcare provider.

SUMMARY:
The purpose of this Expanded Access Program (EAP) is to allow patients to continue receiving treatment with copanlisib if they are currently having, in the opinion of their healthcare provider, an objective favorable response when taking copanlisib. Patients considering this access program should have no other therapeutic option, have not developed a disease and/or medical condition (including pregnancy), and/or have a toxicity that would conflict with continuing to receive copanlisib.

ELIGIBILITY:
Inclusion Criteria:

* Patient has provided written informed consent.
* Patient meets one of the following criteria:

  * Already enrolled and on treatment with copanlisib in Bayer-sponsored Study 17067 (CHRONOS-3), OR
  * Already enrolled and on treatment with copanlisib in an investigator-initiated research (IIR)/institution-sponsored collaborative study (ISCS), OR
  * Currently on copanlisib treatment prescribed by a healthcare provider.
* Patient is deriving an objective favorable response from copanlisib in the opinion of their healthcare provider.
* Patient has no suitable alternative treatments available.
* Women of childbearing potential and men must agree to use effective contraception when sexually active due to potential embryo-fetal toxicity for 1 month after the last dose.

Exclusion Criteria:

* Patients who may have developed a disease/condition/toxicity that would conflict with continuing to receive copanlisib treatment.
* Patients on treatment with rituximab (R) either alone or in combination with chemotherapy, including an alkylating agent (e.g. bendamustine [R-B] or cyclophosphamide, hydroxydoxorubicin, vincristine, prednisone [R-CHOP]) for relapsed indolent non-Hodgkin's lymphoma (iNHL).

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (11):
- Many Locations, Multiple Locations, Brazil
- Many Locations, Multiple Locations, Chile
- Many Locations, Multiple Locations, Hong Kong
- Many Locations, Multiple Locations, Hungary
- Many Locations, Multiple Locations, Ireland
- Many Locations, Multiple Locations, Malaysia
- Many Locations, Multiple Locations, Poland
- Many Locations, Multiple Locations, Romania
- Many Locations, Multiple Locations, Russia
- Many Locations, Multiple Locations, Taiwan
- Many Locations, Multiple Locations, Ukraine